CLINICAL TRIAL: NCT06032403
Title: Patient with Atopic Dermatitis' Needs for Self-management Support - Flexible Patient Centred Consultations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Aage Bangs Fond (Other); The Novo Nordic Foundation (Other); Herlev and Gentofte Hospital (Other); Sanofi (Industry); Almirall, S.A. (Industry)
Responsible Party: Principal Investigator, Anna Sophie Belling Krontoft, Clinical Nurse specialist at the Department of Dermatology and Allergy, Principal investigator and PhD student, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: UHGentofte P-2022-298; H-22048513 (Other: The National Committee on Health Research Ethics)
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis
Keywords: Patient-centred care; Self-management support
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: The investigators start by including 100 participants (control group) who are attending the clinical. The control group will be followed for one year. After the control group has been followed for one year the investigators include 100 participants in the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Consists of 100 participants followed for one year
- Intervention group (Other): Consists of 100 participants followed for one year
  Interventions: Behavioral: flexible patient centred consultations

INTERVENTIONS:
Behavioral: flexible patient centred consultations — In the intervention group, the set-up will be flexible patient-centred consultations. The first consultation for the participant will be with the doctor and depending on the participant's need, the following consultations can be scheduled as either a doctor- or a nurse consultation. After each consultation, it will be decided in collaboration between the healthcare professionals and the participant whether a nurse or a doctor consultation will be relevant next. The consultations (whether it is with the doctor or nurse) will be centered around the participant's choice of topics by use of an atopic dermatitis dialogue tool developed in the department. Additionally, the nurse consultation will focus on therapeutic patient education (TPE) in atopic dermatitis. The interval between consultations will depend on the participant's need
  Arms: Intervention group

SUMMARY:
In this study, the investigators will conduct a controlled trial to investigate the effects of a flexible patient-centred consultation with a focus on self-management support, well-being, treatment content, and self-management skills in patients with atopic dermatitis.

The investigators will include 200 participants; 100 participants in a control group followed by 100 participants in an intervention group. The controlled trial will take place at the outpatient clinic at the Department of Dermatology and Allergy, Herlev-Gentofte Hospital and the daily management will be done by the project manager/Ph.d. student with support from the project group.

In the control group, participants will be provided with care as usual. This means participants will be seen by a doctor and new participants will get an additional nurse session focusing on therapeutic patient education (TPE) in atopic dermatitis. The consultations are scheduled at regular intervals of approximately three months but with alterations if the participant needs to be seen before.

In the intervention group, the set-up will be flexible patient-centred consultations. The first consultation for the participant will be with the doctor and depending on the participant's need, the following consultations can be scheduled with either a doctor- or a nurse consultation. After each consultation, it will be decided in collaboration between the healthcare professionals and the participant whether a nurse or a doctor consultation will be relevant next. The consultations (whether it is with the doctor or nurse) will be centered around the participant's choice of topics by use of an atopic dermatitis dialogue tool developed in the department. Additionally, the nurse consultation will focus on therapeutic patient education (TPE) in atopic dermatitis. The interval between consultations will depend on the participant's need

DETAILED DESCRIPTION:
In this study, the investigators will conduct a controlled trial to investigate the effects of a flexible patient-centred consultation with a focus on self-management support, well-being, treatment content, and self-management skills in patients with atopic dermatitis.

The investigators will include 200 participants; 100 participants in a control group followed by 100 participants in an intervention group. The controlled trial will take place at the outpatient clinic at the Department of Dermatology and Allergy, Herlev-Gentofte Hospital and the daily management will be done by the project manager/Ph.d. student with support from the project group.

In the control group, participants will be provided with care as usual. This means participants will be seen by a doctor and new participants will get an additional nurse session focusing on therapeutic patient education (TPE) in atopic dermatitis. The consultations are scheduled at regular intervals of approximately three months but with alterations if the patients need to be seen before.

In the intervention group, the set-up will be flexible patient-centred consultations. The first consultation for the participant will be with the doctor and depending on the participant's need, the following consultations can be scheduled with either a doctor- or a nurse consultation. After each consultation, it will be decided in collaboration between the healthcare professionals and the participant whether a nurse or a doctor consultation will be relevant next. The consultations (whether it is with the doctor or nurse) will be centered around the participant's choice of topics by use of an atopic dermatitis dialogue tool developed in the department. Additionally, the nurse consultation will focus on therapeutic patient education (TPE) in atopic dermatitis. The interval between consultations will depend on the patient's need

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of atopic atopic dermatitis
* Children and adolescents under 18 years
* Adults over 18 years
* Need to be followed at the department
* Patient or caregiver must be able to speak and understand Danish
* Received oral and written information
* The patient or caregiver has signed the informed consent

Exclusion Criteria:

* A person deprived of liberty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The Well-Being Index (WHO-5) | baseline, 6 and 12 months
  Well-Being Index: WHO-5. WHO-5 is validated for adults and children down to 10-years-old, but as research state that the whole family is affected by the burden of a child's atopic dermatitis, the parent attending a consultation with a child at or under 10 years old will be asked to answer the WHO-5 according to how they believe the participant are feeling. The WHO-5 contains of five statements and a response scale that goes from 0-5 (five representing the highest positive well-being for the participant).
  Points from each question are added together and the sum is multiplied by 4. That will give a number between 0-100. The higher sum score the better the well-being.

SECONDARY OUTCOMES:
The Infant Dermatology Life Quality Index (IDLQI) | baseline, 6 and 12 months
  The Infant Dermatology Quality of Life Index contains 10 questions and a response scale divided into four boxes. Each box gives a point between 0 and 3. The lower number is understood as the most positive for the participant.
  The index is filled out by a parent to a participating child between the ages of 0 to 5 years.
  Points from each question are added together and the end-sum represents the score. The sum score can be between 0 and 30. The higher the score the worse the assumed quality of life.
The Dermatology Life Quality Index (DLQI) | baseline, 6 and 12 months
  The Dermatology Life Quality Index contains 10 questions and a response scale divided into four boxes. Each box gives a point between 0 and 3. The lower number is understood as the most positive for the participant.
  The index is filled out by participants over the age of 15 years.
  Points from each question are added together and the end-sum represents the score. The sum score can be between 0 and 30. The higher the score the worse the assumed quality of life.
The Children Dermatology Life Quality Index (CDLQI) | baseline, 6 and 12 months
  The Children Dermatology Life Quality Index contains 10 questions and a response scale divided into four boxes. Each box gives a point between 0 and 3. The lower number is understood as the most positive for the participant.
  Question number 7 is only applicable if the participant is attending school.
  The index is filled out by participants (a parent when the participant is between 5 and 10 years old and the participant themselves when the participant is between 10-15 years old).
  Points from each question are added together and the end-sum represents the score. The sum score can be between 0 and 30. The higher the score the worse the assumed quality of life
The Patient Oriented eczema measure (POEM) | baseline, 6 and 12 months
  A subjective patient measure of eczema severity.
  The questionnaire contains 7 questions and a response scale with 5 options. Each option gives a point between 0 and 4. The sum score is found by adding the points together. The sum score can be between 0-28. The higher the sum score the worse the assumed severity of eczema.
  The questionnaire is filled out by participants over the age of 15 years.
The Patient Oriented eczema measure for parents (POEM for parents) | baseline, 6 and 12 months
  A subjective patient measure of eczema severity.
  The questionnaire contains 7 questions and a response scale with 5 options. Each option gives a point between 0 and 4. The sum score is found by adding the points together. The sum score can be between 0-28. The higher the sum score the worse the assumed severity of eczema.
  The questionnaire is filled out by a parent to a participant under the age of 10 years and together with the participant if the participant is between 10 and 15 years old.
Eczema And Severity Index (EASI) | baseline, 6 and 12 months
  Assessment of eczema severity. Filled out by healthcare professionals at consultation visits.
  The EASI contains of a severity score between 0-3 and an area score between 0-6. These scores are given for each of the four body regions (head and neck, trunk, over-extremities, and under-extremities). The minimum EASI score is 0 and the maximum EASI score is 72. The higher the sum-score the worse the eczema severity.
Pruritus numeric rating scale (Pruritus NRS). | baseline, 6 and 12 months
  Scale for measuring itch. Consists of a horizontal line with 11 boxes going from 0 to 10 (from left to right). 0 being no itch and 10 being the worst imaginable itch. The scale is answered two times first thinking about the last 24 hours and secondly thinking about an average over the last 7 days. The sum-score for is calculated for each question and can be between 0 and 10. The higher the score the worse the pruritus is.
  The scale is filled out by participants over the age of 15 years. By a parent together with the participant if the participant is between 10-15 years old. By a parent to a participant if the participant is under 10 years old.
The sleep disturbance numeric rating scale (SD NRS) | baseline, 6 and 12 months
  Scale for measuring sleep disturbance. Consists of a horizontal line with 11 boxes going from 0 to ten (from left to right). 0 being no sleep disturbance and 10 being I can´t sleep at all. The scale is answered two times first thinking about the last 24 hours and secondly thinking about an average over the last 7 days. The sum-score is calculated for each question and can be between 0 and 10. The higher the score the worse the sleep disturbance is considered.
  The scale is filled out by participants over the age of 15 years. By a parent together with the participant if the participant is between 10-15 years old. By a parent to a participant if the participant is under 10 years old.
Patient activity measures (PAM) | baseline, 6 and 12 months
  For measuring patient activation (self-management). The scale consists of 13 questions with a response scale of 5 boxes (highly disagree, disagree, agree, very much agree, and don't know). Each answer corresponds to a point between 0-4.
  The raw sum score is done by adding each point and dividing the point total by the number of items completed with a 1-4. and then multiply by 13. Secondly, the investigators convert the raw score into the activation score by using the "Insignia health License package". The activation score can be between 0 and 100. The higher the score the less patient activity in regards to the disease (atopic dermatitis).
  The PAM is filled out by participants over 15 years of age
Questionnaire about patient and healthcare collaboration (CollaboRATE) | baseline, 6 and 12 months
  Scale for measuring involvement of the patient in the consultation. The scale consist of three questions each with a response scale going from 0-9 (0 = not at all and 9 = to a high degree). The sum score is done by adding the points from each question. The sum score can be between 0-27. The higher the score the better the assumed involvement of the patient in the consultation.

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte University Hospital, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No